CLINICAL TRIAL: NCT01943383
Title: PHARMACOGENOMIC EVALUATION OF ANTIHYPERTENSIVE RESPONSES IN INDUCED PLURIPOTENT STEM (IPS) CELLS STUDY (PEAR-IPSC) (PEAR-iPSC)
Brief Title: Pharmacogenomic Evaluation of Antihypertensive Responses in Induced Pluripotent Stem (iPS) Cells Study
Acronym: PEAR-iPSC
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600901; 093-2013 (Other: IRB)
Record Dates: First submitted 2013-08-27; First posted 2013-09-17 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Induced Pluripotent Stem Cells (iPS cells)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diuretic: Patients who received a diuretic drug during the parent trial are eligible for participation.
  Interventions: Genetic: iPSC

INTERVENTIONS:
Genetic: iPSC — Single blood draw for the production of induced pluripotent stem cells.

SUMMARY:
Patients enrolled in this study will have completed one of the parent studies "Pharmacogenomic Evaluation of Antihypertensive Responses" (PEAR-1 or PEAR-2) evaluating how well their blood pressure was controlled by medication. Patients in the current study will provide a single tube of blood which will be used to create adult stem cells that can be converted into other cell types, like heart or vasculature. Patients will not be asked to return for any follow up visits.

DETAILED DESCRIPTION:
If the patient decide to participate in this study, they will have 1 visit for the study that will include a blood draw. Upon arrival to the clinic, the study will be explained to the patient in detail. The patient will be asked at that time to sign this consent form. The patient will have the opportunity to ask questions and the research staff will answer those questions. If the patient decides to participate in this study and sign a consent form, then a blood sample will be collected from a vein in the arm. A total of 2 teaspoons full of blood will be drawn for the study.

During this visit, in addition to collecting a blood sample, patients will be asked about their medical history and medications they are currently taking, and will have their vital signs assessed, including blood pressure, pulse, and temperature.

Blood will be drawn by a trained nurse or a phlebotomist at a family medicine clinic in Gainesville, Florida. The blood sample will be further processed in laboratories at the University of Florida, for the establishment of iPS cells. iPS cells will retain the patient's genetic makeup which makes them useful for research. Several experiments will be conducted on these cells that will provide data that can be used to learn more about how genetic markers can lead to differences in blood pressure response to medicines. These cells will be used for up to 8 years.

ELIGIBILITY:
Inclusion Criteria:

* participation in the parent trial PEAR (201-2005) or PEAR2 (271-2010)
* assigned to a diuretic arm

Exclusion Criteria:

* no participation in the parent trial PEAR (201-2005) or PEAR2 (271-2010)
* assigned to a beta blocker arm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants recruited from the Pharmacogenomic Evaluation of Antihypertensive Responses studies; PEAR (#201-2005) and PEAR-2 (#271-2010) funded by the National Institutes of Health. Participants in the study have completed either PEAR or PEAR-2 studies
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Cellular gene expression, cellular protein expression, and site directed mutagenesis of induced pluripotent stem cells in response to antihypertensive drugs. | 8 years
  iPSC cells will be used to model the mechanisms by which genetic differences influence responses to antihypertensive drugs. Potential methods included cellular gene expression, cellular protein expression, and site directed mutagenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Johnson, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States